CLINICAL TRIAL: NCT00006290
Title: Perceived Changes in Body Habitus and Body Image Among HIV+ Persons Currently Receiving or Recently Discontinuing Combination Antiretroviral Therapy
Brief Title: Perceived Changes in Body Build and Image in Patients Who Are Now Taking or Recently Have Stopped Taking Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5089; AACTG A5089
Record Dates: First submitted 2000-09-21; First posted 2001-08-31 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Drug Therapy, Combination; Questionnaires; Quality of Life; Patient Compliance; Body Composition; Anti-HIV Agents; Adipose Tissue; Body Image
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Patient Compliance

SUMMARY:
The purpose of this study is to learn how changes in body build affect the lives of people taking anti-HIV medications. By learning this, a set of questions can be created to help understand how changes in body build and image affect people living with HIV infection.

A set of questions used to measure body image might be useful in future HIV studies. It may help doctors understand patient concerns about their body image and why some patients stop taking their anti-HIV medications.

DETAILED DESCRIPTION:
A valid measure of body image would be useful for AACTG studies. Such a measure might permit investigators to examine dissatisfaction with body image as a predictor variable in analyses of premature study drug discontinuation, loss to follow-up, and study drug non-adherence, and as a secondary outcome in antiretroviral and fat redistribution treatment trials.

Six focus group interviews, each lasting approximately 2 hours, are conducted at 4 AACTG sites. Separate groups are run for men and women, and male groups are segmented by sexual orientation. A moderator leads discussions about patients' perceived changes in body habitus and body image. Group interviews are audio-taped and transcribed verbatim. Qualitative interview data are sent electronically to the Data Management Center, where they are thematically analyzed using qualitative data analysis (content analysis) techniques. Salient focus group findings are used to construct questionnaire items.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 18 years or older.
* Are HIV-positive.
* Are experiencing at least 1 of the following symptoms associated with fat changes due to HIV: 1) increase in belt or waist size; 2) increase in size of back of neck; 3) increase in bra, shirt, or blouse size to fit increasing breast size; 4) fat increase in other areas of the body; 5) loss of facial fat; 6) loss of fat in arms or legs; 7) loss of fat in buttocks.
* Agree to protect the confidentiality of other focus group participants.
* Are able to speak and read English.
* Have taken 2 or more anti-HIV medications for a total of at least 6 months at any time before entering this study. Patients must have taken some anti-HIV treatment during the 6-month period before study entry. Patients who have stopped taking these medications in the 6 months before study entry may still be eligible.
* Are willing to talk about personal topics in a taped group interview.
* Are male and either gay or bisexual (if enrolling in the Ohio State University or University of California focus groups).
* Are either female or heterosexual male (if enrolling in the University of Pennsylvania or Johns Hopkins University focus groups).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a mental disability that, in the opinion of the researcher, could interfere with study participation.
* Have already taken part in an A5089 focus group interview.
* Have diabetes or Cushing's disease or have had surgery that might otherwise explain changes in body fat.
* Have changes in diet or physical activity that might explain changes in body fat.
* Have been on glucocorticoid therapy for a long time.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Judith Neidig, Study Chair; William Holmes, Study Chair
Locations (4):
- United States (4):
  - Univ of California, San Diego, San Diego, California
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania